CLINICAL TRIAL: NCT03907020
Title: Application of the Indicator Amino Acid Oxidation Technique for the Determination of Metabolic Availability of Lysine From Barley and Oatmeal Protein, in Young Adult Men
Brief Title: Metabolic Availability of Lysine From Barley in Young Adult Men
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Glenda Courtney-Martin, Dietitian, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1000060245
Record Dates: First submitted 2019-04-05; First posted 2019-04-08 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Meabolic Availabiliy of Barley (Experimental): Healthy adult men
  Interventions: Dietary Supplement: Barley

INTERVENTIONS:
Dietary Supplement: Barley — Assessing the metabolic availability of lysine in barley.

SUMMARY:
Protein is the key determinant of growth and bodily functions. The quality of food proteins depend on their amino acid content and the amount of amino acids used by the body to make proteins. Globally Cereal Grains (CG) provide 50% of the calories and protein in the diet and exceed 80% in poorer developing countries. Barley is an important cereal grain in the diet. The protein in barley is low in the essential amino acid lysine. Hence barley protein is of low quality. Low lysine affects protein synthesis in the body. Cooking methods also affect the lysine available from foods to the body. It is important to assess the effect of different cooking methods on the lysine availability of barley.

DETAILED DESCRIPTION:
Each subjects will receive each of up to 10 experimental diets for the Barley Study (4 reference protein diets providing, 3 Barley diets using dry cooking method, and 3 Barley diets using moist heat cooking method) in random order over a series of up to 10 experimental periods. The reference protein diet will be patterned after the AA pattern of egg protein using crystalline AA as the protein source. Three of the 4 lysine levels will be replaced by lysine provided in Barley each cooked using two different cooking methods ( dry and moist-heat).Each experiment will be conducted over 3 days.

Adaptation days:

During days 1 and 2 the subjects will be adapted to the level of lysine being studied, consuming the same diet as they will receive on day 3 (IAAO study day). The adaptation diet will be consumed as 4 equal meals.Meals will be divided into 4 equal parts to be spread evenly throughout the day and consumed in their usual environment on their usual activities of daily living.

IAAO study day/isotope delivery and sample collection day:

On the oxidation study day 3, following a 12-h overnight fast, subjects will come to the Hospital for Sick Children, Toronto, ON for a period of 5.5 h. On the oxidation study day, the diet is consumed as 9 iso-nitrogenous and iso-energetic hourly meals. Between meals, subjects are allowed to rest on bed, watch television or use a computer. Study days for each participant will be separated by ≥ 1 week. For the duration of all experiments, subjects will consume a daily multivitamin (Centrum Forte, Whitehall Robins) and 500 mg choline supplement (Nature's Way or equivalent), to ensure adequate vitamin intake. The multi vitamin supplement is provided to ensure that no vitamin cofactors are limiting in the diet which could alter metabolic pathways and functioning.

ELIGIBILITY:
Inclusion Criteria:

* Male, age 18 - 40 years, Healthy with no known clinical condition which would affect protein or AA metabolism, ex. Diabetes,
* Stable Body Weight (±0 to 5lb weight gain or loss in the last 3 months)
* Not on any medications that could affect protein or amino acid metabolism e.g. steroids.

Exclusion Criteria:

* Unwillingness to participate or unable to tolerate the diet
* Recent history of weight loss within the last 3 months or on a weight reducing diet Inability to tolerate study diets (ex. Allergy to ingredients).

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Phenylalanine Oxidation | 8 hrs
  Breath samples will be collected from each subject on each study day and the 13C enrichment measured by mass spectrometry. This will be plotted against phenylalanine intake in the reference and barley diets to determine the amount of lysine available in barley.

CONTACTS AND LOCATIONS:
Overall Officials: Glenda Courtney-Martin, PhD, Principal Investigator — Associate Scientist
Locations (1):
- The Hospital For Sick Children, Toronto, Ontario, Canada